CLINICAL TRIAL: NCT02117297
Title: Allogeneic Stem Cell Transplantation Following by Targeted Immune Therapy) (Gemtuzumab Ozogamicin) in Average Risk Acute Myelogenous Leukemia and Myelodysplastic Syndrome (AML/MDS)
Brief Title: SCT Plus Immune Therapy in Average Risk AML/MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Mitchell Cairo, Principal Investigator, New York Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC-504; L 10,394 (Other: New York Medical College)
Record Dates: First submitted 2014-04-08; First posted 2014-04-17 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gemtuzumab Ozogamicin (Experimental): Consolidation therapy with GO will be administered between days 60 and 180 post transplantation when the ANC is >1000/mm3 and platelet count is >40,000/mm3 untransfused x 3 days after AlloSCT and again at minimum 8 weeks later.
  Interventions: Drug: Gemtuzumab Ozogamicin

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin — Gemtuzumab, 9.0 mg/m2, will be given IV over 2 hours two times post allogeneic transplantation.
  Other Names: Mylotarg

SUMMARY:
Allogeneic stem cell transplantation followed by targeted immune therapy with Gemtuzumab Ozogamicin (Mylotarg) will be given to patients with average risk AML or MDS.

DETAILED DESCRIPTION:
Reduced intensity conditioning regimen of Busulfan (Bu) and Fludarabine (Flu) + Anti-Thymocyte Globulin (ATG ) (unrelated donors only) or reduced toxicity conditioning regimen of Bu/Flu/alemtuzumab, or reduced hepatic toxicity regimen of melphan/Flu/alemtuzumab and AlloSCT, followed by Gemtuzumab Ozogamicin consolidation in patients with average risk AML/MDS meeting eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

Disease Status:

* AML 1st CR with a matched family donor
* AML 1st CR with unrelated donor
* AML 2nd CR or CRP
* MDS and < or = 5% bone marrow myeloblasts at diagnosis

Disease Immunophenotype:

* Disease must express a minimum of > or = 10% CD33 positivity for patients with AML

Organ Function:

* Adequate renal function, adequate liver function, adequate cardiac function, adequate pulmonary function

Exclusion Criteria:

* Patients with active CNS AML disease at time of preparative regimen
* Secondary MDS
* Poor cytogenetics
* Female patients who are pregnant
* Karnofsky <70% or Lansky <50% if 10 years or less
* Age >25 years
* Seropositive for HIV

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2012-01-12 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
to evaluate incidence of graft failure | Day +42
  If three or more of the first ten patients experience primary or secondary graft failure, we will discontinue the study.
to evaluate survival rates | 1 year
  Event-free survival and overall survival after RI AlloSCT and targeted immunotherapy in patients with average risk AML/MDS.
to determine toxicity | 1 year
  to monitor for serious adverse events related to protocol investigational therapy

SECONDARY OUTCOMES:
Minor histocompatibility antigen | 1 year
  To measure the minor histocompatibility antigen expression on AML tissue, donor and recipient, and the development of MHA specific CTLs post AlloSCT.
Chimerism | 1 year
  To determine the degree of mixed/complete donor chimerism after RI AlloSCT in patients with average risk AML/MDS.
Graft-versus-host disease | 1 Year
  To estimate the risk of acute and chronic GVHD following RI AlloSCT and FK506/MMF GVHD prophylaxis in patients with average risk AML/MDS.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S. Cairo, M.D., Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided